CLINICAL TRIAL: NCT06119087
Title: Mechanical Insufflation in the Philadelphia Amyotrophic Lateral Sclerosis Cohort (MI-PALS) Study
Acronym: MI-PALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 854981
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Chronic Respiratory Failure; Airway Clearance Impairment; Neuromuscular Diseases
Keywords: amyotrophic lateral sclerosis; chronic respiratory failure; neuromuscular weakness; mechanical insufflation-exsufflation; peak cough flow
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: single-center, single-arm feasibility pilot study of in 20 patients with ALS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mechanical insufflation (Experimental): Participants will be asked to perform mechanical insufflation using the BiWaze cough device as 5 sets of 5 insufflations twice daily for 6 months.
  Interventions: Device: Mechanical insufflation

INTERVENTIONS:
Device: Mechanical insufflation — Mechanical insufflation (MI) is a chest physiotherapy exercise that will be performed using a type of mechanical insufflator-exsufflator (MI-E) known as the BiWaze Cough device. The device connects to a tube that can interface with a patient using either a facemask or mouthpiece.
  Mechanical insufflation is a chest physiotherapy exercise that passively inflates the chest with positive pressure that is delivered in coordination with the patient's own inspiratory timing until maximal inflation capacity (MIC), determined by the patient or maximal chest rise on visual inspection. At MIC, the patient passively exhales, which completes one "cycle". Prior literature has used a "dose" of 5 sets of 5 cycles once or twice daily. The maneuver is usually performed with assistance of a caregiver to hold the mask or mouthpiece in place.

SUMMARY:
The goal of this clinical trial is to learn how doing mechanical insufflation (MI) using a mechanical insufflator-exsufflator (MI-E) device affects breathing in early amyotrophic lateral sclerosis (ALS). This will be a single-center, single-arm study of MI in 20 patients with ALS at Penn.

Based on prior research, we believe that 6-months of MI may slow decline in cough strength, measured as peak cough flow (PCF).

Participants will perform MI using a device designed for mechanical insufflation-exsufflation (MI-E) known as the BiWaze Cough system. The BiWaze Cough is used for mucus clearance . It is connected to tubing and mouthpiece (or mask). The device will use programmed pressure and timing settings. An insufflation includes inflating the lungs for a maximal size inhalation before exhaling. The daily routine for the device includes 5 sets of 5 insufflations twice daily.

Researchers will compare how use of MI in early ALS affects peak cough flow compared to 20 subjects who did not use MI in early ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age ≥18 years.
4. Diagnosed with amyotrophic lateral sclerosis using the Gold Coast Criteria.
5. Have an able and willing caregiver to assist with mechanical insufflation on a daily basis.
6. Willingness and ability to participate in study procedures.

Exclusion Criteria:

1. Age <18 years old.
2. Inability to perform a cough peak flow or spirometry manuever
3. Current use of non-invasive ventilation (NIV), bi-level positive pressure ventilation, or "Bi-PAP" or physician prescribing NIV on day of potential enrollment.
4. Current use of MI-E (also known as a "cough assist device") for airway clearance. Please note that patients can start use of a MI-E device subsequent to enrollment while currently being followed for the study.
5. Active enrollment in hospice.
6. Current tracheostomy.
7. Presence of cognitive dysfunction that would impair ability to complete study procedures, as determined by neurology attending physician.
8. Absence of an able and willing caregiver to assist with MI twice daily as specified in the protocol.
9. Pregnancy
10. Medical history of any of the following:

    1. Recent hemoptysis
    2. Recent barotrauma
    3. History of emphysema of any kind (including bullous emphysema)
    4. History of or known susceptibility to pneumothorax
    5. History of or known susceptibility to pneumomediastinum
    6. Chronic obstructive pulmonary disease
    7. Uncontrolled asthma (defined as recent exacerbation requiring corticosteroids in the previous 30 days)
    8. Symptomatic cardiomyopathy (heart failure) with left ventricular ejection fraction less than 50%
    9. History of right heart failure or pulmonary hypertension
11. Current smoker or tobacco use within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
peak cough flow (PCF) | 6 months
  PCF in liters/minute as measured by use of a peak flow meter while the patient is in a seated upright position. An alternative device for measuring PCF can be the use of a handheld spirometer and using the measured peak expiratory flow by multiplying by 60 to convert from liters/second to liters/minute.
  The subject must be seated in an upright position and the interface must include a mouthpiece or an oronasal mask. Subjects are asked to perform a deep inhalation followed by a maximal cough.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 6 months
  Defined as maximal volume, in liters, that a person can exhale forcefully after a complete inhalation.
  Measured using a spirometer connected to a face mask or mouthpiece in the sitting and upright position.
Maximal inspiratory pressure (MIP) | 6 months
  Defined as the maximum pressure, in cmH2O, generated when the subject exhales as much air as possible and then immediately inhales as forcefully as possible.
Maximal expiratory pressure (MEP) | 6 months
  Defined as the maximum pressure, in cmH2O, generated when the subject inhales as much air as possible and then immediately exhales as forcefully as possible.
  Measured using a hand-held manual or digital manometer connected to a mouthpiece or mask in the sitting and upright position.
Maximum insufflation capacity (MIC) | 6 months
  Defined as exhaled volume, in liters, immediately following a MI maneuver to maximum insufflation capacity.
  Measured using a spirometer connected to a face mask or mouthpiece, in the sitting and upright position.
Maximum insufflation capacity assisted peak cough flow | 6 months
  Defined as the peak cough flow generated from MIC.
  Lungs are inflated to MIC using MI and before the subject exhales they insert a peak flow meter in their mouth and follow with a peak cough flow as described above.
MIC-FVC difference | 6 months
  defined by subtracting the FVC from the MIC
Transcutaneous carbon dioxide | 6 months
  Defined as the average value in mmHg from a daytime in-clinic measurement over a 15-minute transcutaneous recording.
  Measured using a Sentec transcutaneous digital monitoring system while the subject is sitting upright in a chair or wheelchair. The transcutaneous sensor can be placed on the subject forehead, cheek, or earlobe.
ALS Functional Rating Scale - Revised (ALSFRS-R) dyspnea and orthopnea scores | 6 months
  The ALSFRS-R is a 12-item standardized questionnaire to assess the motor function status of an individual with ALS. The ALSFRS-R is assessed by a research staff member who has been certified for performance of the ALSFRS-R.
  The dyspnea score is one of the questions focusing on level of shortness of breath, scored on a scale of 0 to 4, with 4 being no symptoms at all and 0 being severely symptomatic with consideration of mechanical respiratory support.
  The orthopnea score is one of the questions focused on breathing symptoms and difficulty sleeping while lying supine, scored on a scale of 0 to 4, with 4 being no symptoms at all and 0 being severely symptomatic with inability to sleep.
Global rate of change score for peak cough flow | 6 months
  The global rate of change score for the peak cough flow will ask patients how effective they think their cough is today by rating it on a Likert scale from -7 (extremely impaired) to +7 (extremely strong).

OTHER OUTCOMES:
Time to start of non-invasive ventilation | 1 year
  Defined by the time period between enrollment for the MI trial and date of prescription for non-invasive ventilation
  Non-invasive ventilation start date will be defined by date of prescription for non-invasive ventilation as recorded in the medical record or patient-reported date if a prescription is not recorded in the medical record.
Tracheostomy free survival time | 1 year
  Defined by the time period between enrollment for the MI trial and death as long as the subject never had a tracheostomy placed.
  Death date will be determined by family report, electronic medical record review, or publicly available obituaries.
  Tracheostomy placement will be determined by patient or family report; or as documented in the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ackrivo, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaminska M, Browman F, Trojan DA, Genge A, Benedetti A, Petrof BJ. Feasibility of Lung Volume Recruitment in Early Neuromuscular Weakness: A Comparison Between Amyotrophic Lateral Sclerosis, Myotonic Dystrophy, and Postpolio Syndrome. PM R. 2015 Jul;7(7):677-684. doi: 10.1016/j.pmrj.2015.04.001. Epub 2015 Apr 3. PMID 25845857
- [Background] Katz SL, Barrowman N, Monsour A, Su S, Hoey L, McKim D. Long-Term Effects of Lung Volume Recruitment on Maximal Inspiratory Capacity and Vital Capacity in Duchenne Muscular Dystrophy. Ann Am Thorac Soc. 2016 Feb;13(2):217-22. doi: 10.1513/AnnalsATS.201507-475BC. PMID 26599476
- [Background] McKim DA, Katz SL, Barrowman N, Ni A, LeBlanc C. Lung volume recruitment slows pulmonary function decline in Duchenne muscular dystrophy. Arch Phys Med Rehabil. 2012 Jul;93(7):1117-22. doi: 10.1016/j.apmr.2012.02.024. Epub 2012 Mar 12. PMID 22421625
- [Background] Chiou M, Bach JR, Jethani L, Gallagher MF. Active lung volume recruitment to preserve vital capacity in Duchenne muscular dystrophy. J Rehabil Med. 2017 Jan 19;49(1):49-53. doi: 10.2340/16501977-2144. PMID 27630091
- [Background] Mustfa N, Aiello M, Lyall RA, Nikoletou D, Olivieri D, Leigh PN, Davidson AC, Polkey MI, Moxham J. Cough augmentation in amyotrophic lateral sclerosis. Neurology. 2003 Nov 11;61(9):1285-7. doi: 10.1212/01.wnl.0000092018.56823.02. PMID 14610141
- [Background] Chatwin M, Bush A, Simonds AK. Outcome of goal-directed non-invasive ventilation and mechanical insufflation/exsufflation in spinal muscular atrophy type I. Arch Dis Child. 2011 May;96(5):426-32. doi: 10.1136/adc.2009.177832. Epub 2010 Jun 23. PMID 20573738
- [Background] Vianello A, Corrado A, Arcaro G, Gallan F, Ori C, Minuzzo M, Bevilacqua M. Mechanical insufflation-exsufflation improves outcomes for neuromuscular disease patients with respiratory tract infections. Am J Phys Med Rehabil. 2005 Feb;84(2):83-8; discussion 89-91. doi: 10.1097/01.phm.0000151941.97266.96. PMID 15668554
- [Background] Miske LJ, Hickey EM, Kolb SM, Weiner DJ, Panitch HB. Use of the mechanical in-exsufflator in pediatric patients with neuromuscular disease and impaired cough. Chest. 2004 Apr;125(4):1406-12. doi: 10.1378/chest.125.4.1406. PMID 15078753
- [Background] Tzeng AC, Bach JR. Prevention of pulmonary morbidity for patients with neuromuscular disease. Chest. 2000 Nov;118(5):1390-6. doi: 10.1378/chest.118.5.1390. PMID 11083691
- [Background] Bach JR, Goncalves MR, Hamdani I, Winck JC. Extubation of patients with neuromuscular weakness: a new management paradigm. Chest. 2010 May;137(5):1033-9. doi: 10.1378/chest.09-2144. Epub 2009 Dec 29. PMID 20040608
- [Background] Vitacca M, Paneroni M, Trainini D, Bianchi L, Assoni G, Saleri M, Gile S, Winck JC, Goncalves MR. At home and on demand mechanical cough assistance program for patients with amyotrophic lateral sclerosis. Am J Phys Med Rehabil. 2010 May;89(5):401-6. doi: 10.1097/PHM.0b013e3181d89760. PMID 20407305
- [Background] Chatwin M, Toussaint M, Goncalves MR, Sheers N, Mellies U, Gonzales-Bermejo J, Sancho J, Fauroux B, Andersen T, Hov B, Nygren-Bonnier M, Lacombe M, Pernet K, Kampelmacher M, Devaux C, Kinnett K, Sheehan D, Rao F, Villanova M, Berlowitz D, Morrow BM. Airway clearance techniques in neuromuscular disorders: A state of the art review. Respir Med. 2018 Mar;136:98-110. doi: 10.1016/j.rmed.2018.01.012. Epub 2018 Feb 6. PMID 29501255
- [Background] Miller RG, Jackson CE, Kasarskis EJ, England JD, Forshew D, Johnston W, Kalra S, Katz JS, Mitsumoto H, Rosenfeld J, Shoesmith C, Strong MJ, Woolley SC; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter update: the care of the patient with amyotrophic lateral sclerosis: drug, nutritional, and respiratory therapies (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2009 Oct 13;73(15):1218-26. doi: 10.1212/WNL.0b013e3181bc0141. PMID 19822872
- [Background] Sawnani H, Mayer OH, Modi AC, Pascoe JE, McConnell K, McDonough JM, Rutkowski AM, Hossain MM, Szczesniak R, Tadesse DG, Schuler CL, Amin R. Randomized trial of lung hyperinflation therapy in children with congenital muscular dystrophy. Pediatr Pulmonol. 2020 Sep;55(9):2471-2478. doi: 10.1002/ppul.24954. Epub 2020 Jul 20. PMID 32658385
- [Background] McDonald LA, Berlowitz DJ, Howard ME, Rautela L, Chao C, Sheers N. Pneumothorax in neuromuscular disease associated with lung volume recruitment and mechanical insufflation-exsufflation. Respirol Case Rep. 2019 Jun 13;7(6):e00447. doi: 10.1002/rcr2.447. eCollection 2019 Aug. PMID 31210952
- [Background] Westermann EJ, Jans M, Gaytant MA, Bach JR, Kampelmacher MJ. Pneumothorax as a complication of lung volume recruitment. J Bras Pneumol. 2013 May-Jun;39(3):382-6. doi: 10.1590/S1806-37132013000300017. PMID 23857693
- [Background] Suri P, Burns SP, Bach JR. Pneumothorax associated with mechanical insufflation-exsufflation and related factors. Am J Phys Med Rehabil. 2008 Nov;87(11):951-5. doi: 10.1097/PHM.0b013e31817c181e. PMID 18617862
- [Background] Cleary S, Misiaszek JE, Kalra S, Wheeler S, Johnston W. The effects of lung volume recruitment on coughing and pulmonary function in patients with ALS. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Mar;14(2):111-5. doi: 10.3109/17482968.2012.720262. Epub 2012 Sep 12. PMID 22970725
- [Background] Cleary S, Misiaszek JE, Wheeler S, Kalra S, Genuis SK, Johnston WS. Lung volume recruitment improves volitional airway clearance in amyotrophic lateral sclerosis. Muscle Nerve. 2021 Dec;64(6):676-682. doi: 10.1002/mus.27417. Epub 2021 Sep 28. PMID 34505708
- [Background] Lechtzin N, Shade D, Clawson L, Wiener CM. Supramaximal inflation improves lung compliance in subjects with amyotrophic lateral sclerosis. Chest. 2006 May;129(5):1322-9. doi: 10.1378/chest.129.5.1322. PMID 16685025
- [Background] Katz SL, Mah JK, McMillan HJ, Campbell C, Bijelic V, Barrowman N, Momoli F, Blinder H, Aaron SD, McAdam LC, Nguyen TTD, Tarnopolsky M, Wensley DF, Zielinski D, Rose L, Sheers N, Berlowitz DJ, Wolfe L, McKim D. Routine lung volume recruitment in boys with Duchenne muscular dystrophy: a randomised clinical trial. Thorax. 2022 Aug;77(8):805-811. doi: 10.1136/thoraxjnl-2021-218196. Epub 2022 Mar 2. PMID 35236763
- [Background] Gomez-Merino E, Bach JR. Duchenne muscular dystrophy: prolongation of life by noninvasive ventilation and mechanically assisted coughing. Am J Phys Med Rehabil. 2002 Jun;81(6):411-5. doi: 10.1097/00002060-200206000-00003. PMID 12023596
- [Background] Bach JR, Baird JS, Plosky D, Navado J, Weaver B. Spinal muscular atrophy type 1: management and outcomes. Pediatr Pulmonol. 2002 Jul;34(1):16-22. doi: 10.1002/ppul.10110. PMID 12112792
- [Background] Bach JR. Amyotrophic lateral sclerosis: prolongation of life by noninvasive respiratory AIDS. Chest. 2002 Jul;122(1):92-8. doi: 10.1378/chest.122.1.92. PMID 12114343
- [Background] Bach JR, Kang SW. Disorders of ventilation : weakness, stiffness, and mobilization. Chest. 2000 Feb;117(2):301-3. doi: 10.1378/chest.117.2.301. No abstract available. PMID 10669664
- [Background] BECK GJ, SCARRONE LA. Physiological effects of exsufflation with negative pressure (E.W.N.P.). Dis Chest. 1956 Jan;29(1):80-95. doi: 10.1378/chest.29.1.80. No abstract available. PMID 13277451
- [Background] Winck JC, Goncalves MR, Lourenco C, Viana P, Almeida J, Bach JR. Effects of mechanical insufflation-exsufflation on respiratory parameters for patients with chronic airway secretion encumbrance. Chest. 2004 Sep;126(3):774-80. doi: 10.1378/chest.126.3.774. PMID 15364756
- [Background] Brinkmann JR, Andres P, Mendoza M, Sanjak M. Guidelines for the use and performance of quantitative outcome measures in ALS clinical trials. J Neurol Sci. 1997 Mar 20;147(1):97-111. doi: 10.1016/s0022-510x(96)05220-3. PMID 9094067
- [Background] Stanojevic S, Kaminsky DA, Miller MR, Thompson B, Aliverti A, Barjaktarevic I, Cooper BG, Culver B, Derom E, Hall GL, Hallstrand TS, Leuppi JD, MacIntyre N, McCormack M, Rosenfeld M, Swenson ER. ERS/ATS technical standard on interpretive strategies for routine lung function tests. Eur Respir J. 2022 Jul 13;60(1):2101499. doi: 10.1183/13993003.01499-2021. Print 2022 Jul. PMID 34949706
- [Background] Shefner JM, Al-Chalabi A, Baker MR, Cui LY, de Carvalho M, Eisen A, Grosskreutz J, Hardiman O, Henderson R, Matamala JM, Mitsumoto H, Paulus W, Simon N, Swash M, Talbot K, Turner MR, Ugawa Y, van den Berg LH, Verdugo R, Vucic S, Kaji R, Burke D, Kiernan MC. A proposal for new diagnostic criteria for ALS. Clin Neurophysiol. 2020 Aug;131(8):1975-1978. doi: 10.1016/j.clinph.2020.04.005. Epub 2020 Apr 19. No abstract available. PMID 32387049
- [Background] Molgat-Seon Y, Hannan LM, Dominelli PB, Peters CM, Fougere RJ, McKim DA, Sheel AW, Road JD. Lung volume recruitment acutely increases respiratory system compliance in individuals with severe respiratory muscle weakness. ERJ Open Res. 2017 Mar 14;3(1):00135-2016. doi: 10.1183/23120541.00135-2016. eCollection 2017 Jan. PMID 28326313
- [Background] Srour N, LeBlanc C, King J, McKim DA. Lung volume recruitment in multiple sclerosis. PLoS One. 2013;8(1):e56676. doi: 10.1371/journal.pone.0056676. Epub 2013 Jan 31. PMID 23383293